CLINICAL TRIAL: NCT06832163
Title: Close Loop Smart Weaning Protocol for Inhaled Nitric Oxide Therapy With PPHN
Brief Title: Close Loop Smart Weaning for INO With PPHN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Close-iNO Study
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn; Inhaled Nitric Oxide
Keywords: Inhaled Nitric Oxide; Persistent Pulmonary Hypertension of the Newborn
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Intervention Model Description: In the initial phase of the study, a total of 10 participants are enrolled in a non-controlled single-group pre-trial.
  The subsequent phase is organized into two distinct groups, each comprising 10 participants, resulting in a total of 20 subjects. The groups are categorized as follows:
  ① The experimental group, which utilizes an intelligent closed-loop offline system operating in a linear decline mode;
  ② The control group, which employs an intelligent closed-loop offline system functioning in a step decline mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhaled Nitric Oxide (iNO), the initial concentration of NO withdrawal is 20ppm. (Experimental): In the initial phase of the study, a total of 10 participants are enrolled in a non-controlled single-group pre-trial.
  The subsequent phase is organized into two distinct groups, each comprising 10 participants, resulting in a total of 20 subjects. The groups are categorized as follows:
  ① The experimental group, which utilizes an intelligent closed-loop offline system operating in a linear decline mode;
  ② The control group, which employs an intelligent closed-loop offline system functioning in a step decline mode.
  Interventions: Device: Nitric Oxide Generation and Delivery System

INTERVENTIONS:
Device: Nitric Oxide Generation and Delivery System — The Nitric Oxide Generation and Delivery System is used to deliver nitric oxide for inhalation therapy into the inspiratory limb of the patient breathing circuit in a way that provides a constant concentration of nitric oxide (NO), as set by the user, to the patient throughout the inspired breath.
  iNO devices with intelligent closed-loop offline function are required to meet the import and discharge standards. The initial concentration of NO withdrawal is 20ppm. In accordance with the withdrawal criteria outlined in the Chinese Guidelines, it is essential to conduct a comprehensive efficacy evaluation prior to initiating withdrawal. Furthermore, the process of inhaled nitric oxide (iNO) evacuation should commence only if specific conditions are satisfied.

SUMMARY:
In contemporary clinical practice concerning the administration of inhaled nitric oxide (iNO) within neonatal intensive care units (NICUs), a stepwise reduction approach is frequently employed in accordance with established neonatal guidelines. Nonetheless, the comparative advantages of a linear reduction strategy-characterized by a gradual decrease in inhalation concentration-over the traditional stepwise method in terms of efficacy and safety have yet to be conclusively established. Furthermore, existing iNO delivery devices necessitate that healthcare professionals manually adjust parameters at intervals dictated by the patient's condition. This reliance on subjective clinical judgment often results in variability and a lack of standardization in the duration of the weaning process. Additionally, the protracted and intricate nature of the weaning procedure considerably heightens the workload for healthcare staff. Importantly, the development of a scientifically grounded, standardized, and real-time feedback mechanism for weaning may enhance clinical outcomes for patients and mitigate the risks associated with inappropriate weaning practices or inconsistent manual interventions. Consequently, this study seeks to leverage the newly introduced "intelligent closed-loop weaning" feature of the latest generation of iNO devices to facilitate automated linear concentration reduction during the weaning process. This innovation aims to alleviate the burden on healthcare personnel while establishing a more standardized and scientifically robust weaning protocol. However, it is noteworthy that there is currently a lack of clinical evidence, both domestically and internationally, regarding the safety and efficacy of this device's weaning protocol, underscoring the urgent need to validate its safety and effectiveness in real-world clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. The administration of inhaled nitric oxide (iNO) has commenced or is anticipated to commence for a duration of 24 hours or more, based on a clinical diagnosis of persistent pulmonary hypertension of the newborn (PPHN);
2. There is a demonstrable positive response to iNO treatment;
3. The iNO delivery system employed is appropriate and meets the conditional requirements, featuring an intelligent closed-loop offline functionality;
4. The guardian or legal representative possesses a comprehensive understanding of the potential benefits and risks associated with participation in this study and has expressed a willingness to consent by signing the informed consent document.

Exclusion Criteria:

1. There are established contraindications associated with the use of nitric oxide, which include the following conditions:

   1. Severe hypoplasia of the left heart or duct-dependent congenital heart disease;
   2. Life-threatening congenital anomalies and congestive heart failure;
   3. Congenital methemoglobinemia;
   4. Significant hemorrhagic events, such as intracranial hemorrhage, intraventricular hemorrhage, and pulmonary hemorrhage.
2. Patients with chronic pulmonary conditions and other refractory diseases are not permitted to initiate withdrawal from the inhaled nitric oxide (iNO) treatment within a seven-day period following its administration.
3. In cases where there is no observable response to iNO or if the duration of use is less than 30 minutes, a strict tapering protocol for withdrawal is not required.
4. If the concentration of iNO treatment exceeds 20 parts per million (ppm) during the initiation phase or if the starting concentration for withdrawal is below 20 ppm, specific considerations must be taken into account.
5. Participation in concurrent clinical trials involving other pharmacological agents or medical devices is prohibited.
6. The investigator may determine that participation in this study is not appropriate for certain individuals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of nitric oxide (NO) rebound hypoxia during the evacuation process | Completion of evacuation (expected day 2 of evacuation)
  The occurrence of nitric oxide (NO) rebound hypoxia during the evacuation process, operationally defined as the frequency of instances in which peripheral capillary oxygen saturation (SpO2) decreased by more than 5% and the fraction of inspired oxygen (FiO2) increased by 15% in order to maintain partial pressure of arterial oxygen (PaO2) above 60 mmHg (with SpO2 ≥ 90%) during the evacuation of NO
The total duration of inhaled nitric oxide (iNO) evacuation | Completion of evacuation (expected day 2 of evacuation)
  The entire length of time required to remove or discontinue the use of iNO.

SECONDARY OUTCOMES:
Device Alarm Frequency | Completion of evacuation (expected day 2 of evacuation)
  The frequency of device alarms recorded during the evacuation process.
NO Concentration Adjustments | Completion of evacuation (expected day 2 of evacuation)
  The total number of adjustments made to knobs and settings for nitric oxide concentration during evacuation.
Mechanical Ventilation Duration | Completion of evacuation (expected day 2 of evacuation)
  The duration of mechanical ventilation.
Adverse Events Incidence | Completion of evacuation (expected day 2 of evacuation)
  The incidence of adverse events associated with nitric oxide treatment.
Complication Rate | Completion of evacuation (expected day 2 of evacuation)
  The complication rate, specifically focusing on Grade 3-4 intraventricular hemorrhage, intraventricular plasmalacia, moderate to severe bronchopulmonary dysplasia, retinopathy of prematurity necessitating intervention, patent ductus arteriosus requiring either medical or surgical management, pulmonary hemorrhage, and air leak syndrome.
ECMO Utilization Rate | Completion of evacuation (expected day 2 of evacuation)
  The proportion of cases that required extracorporeal membrane oxygenation (ECMO).
Mortality Rate Before Discharge | Completion of evacuation (expected day 2 of evacuation)
  The mortality rate prior to discharge.
Healthcare Utilization Preferences | Completion of evacuation (expected day 2 of evacuation)
  Scores obtained from questionnaires assessing preferences for healthcare utilization.The Likert Scale is used in the questionnaires to measure respondents' attitudes, preferences, or perceptions. It typically ranges from 1 to 5 points, where 1 represents "Strongly Disagree" and 5 represents "Strongly Agree". Respondents select the level that best reflects their opinion, allowing researchers to quantify subjective data and analyze trends effectively.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yuan, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No